CLINICAL TRIAL: NCT05169944
Title: A Phase 1 Study of Magrolimab in Children and Adults With Recurrent or Progressive Malignant Brain Tumors
Brief Title: Magrolimab in Children and Adults With Recurrent or Progressive Malignant Brain Tumors
Acronym: PNOC025
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Sabine Mueller, MD, PhD, Principal Investigator, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 210811; NCI-2021-13440 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-12-14; First posted 2021-12-27 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Brain Cancer; Malignant Brain Tumor; Recurrent Brain Tumor; Progressive Malignant Brain Tumor; Brain Tumor, Pediatric; Brain Tumor Adult
Keywords: CD47-signal receptor protein-alpha; Ferumoxytol MRI
MeSH Terms: conditions — Brain Neoplasms | interventions — magrolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Magrolimab) (Experimental): Each participant will receive magrolimab intravenously (IV) at a priming dose of 1 mg/kg during Cycle 0, followed by either 30 mg/kg or 45mg mg/kg dose weekly for eight weeks (Cycles 1 and 2), followed by either 30 mg/kg or 45 mg/kg dose every two weeks for the remainder of the study.
  Interventions: Drug: Magrolimab

INTERVENTIONS:
Drug: Magrolimab — Anti-cancer therapeutic agent targeting the CD47-signal receptor protein-alpha (SIRP-alpha) axis
  Other Names: Anti-CD47 Monoclonal Antibody

SUMMARY:
Children and adults with recurrent or progressive malignant brain tumors have a dismal prognosis, and outcomes remain very poor. Magrolimab is a first-in-class anticancer therapeutic agent targeting the Cluster of differentiation 47 (CD47)-signal receptor protein-alpha (SIRP-alpha) axis. Binding of magrolimab to human CD47 on target malignant cells blocks the "don't eat me" signal to macrophages and enhances tumor cell phagocytosis. Pre-clinical studies have shown that treatment with magrolimab leads to prolonged survival in models of Atypical Teratoid Rhabdoid Tumors (ATRT), diffuse intrinsic pontine glioma (DIPG), high-grade glioma (adult and pediatric), medulloblastoma, and embryonal tumors formerly called Primitive Neuro-Ectodermal Tumors (PNET). Safety studies in humans have proven that magrolimab has an excellent safety profile. Ongoing studies are currently testing magrolimab in adult myelodysplastic syndromes, acute myeloid leukemia, non-Hodgkin lymphoma, colorectal, ovarian, and bladder cancers. Herein we propose to test the safety of magrolimab in children and adults with recurrent or progressive malignant brain tumors.

DETAILED DESCRIPTION:
This is a single arm, 2 strata multi-center study that will be conducted through the Pacific Pediatric Neuro-oncology Consortium (PNOC). Stratum A consists of children (ages 3-17) with recurrent or progressive malignant brain tumors and Stratum B consists of adults (ages ≥ 18) with recurrent or progressive malignant brain tumors. Participants with midline tumors (e.g., midline high grade gliomas (HGG), DIPG, and diffuse midline glioma) will be excluded.

PRIMARY OBJECTIVES:

Children (3-17 years of age)

1. To assess the safety and tolerability of magrolimab in children (Stratum A) with recurrent or progressive malignant brain tumors.
2. To determine the recommended Phase 2 dose (RP2D) for magrolimab in children (Stratum A) with recurrent or progressive malignant brain tumors.

Adults (18 years and older)

1. To assess the safety and tolerability of magrolimab in adults (Stratum B) with recurrent or progressive malignant brain tumors.
2. To determine the recommended Phase 2 dose for magrolimab in adults (Stratum B) with recurrent or progressive malignant brain tumors.

EXPLORATORY OBJECTIVES:

1. To evaluate the pharmacokinetic (PK) profile of magrolimab in blood and cerebrospinal fluid (CSF) in children and adults with recurrent or progressive malignant brain tumors.
2. To evaluate Ferumoxytol MRI imaging as a biomarker for intratumoral macrophages during treatment with magrolimab in children and adults with recurrent or progressive malignant brain tumors.
3. To evaluate the changes in the immune cells in the peripheral blood and CSF and changes in the immune cytokine milieu in the peripheral blood serum and CSF during treatment with magrolimab in children and adults with recurrent or progressive malignant brain tumors.
4. To evaluate the changes in the amounts of cell-free tumor DNA in the peripheral blood and CSF during treatment with magrolimab in children and adults with recurrent or progressive malignant brain tumors.
5. To assess Quality of Life (QOL) and cognitive measures in children and adults with recurrent or progressive malignant brain tumors treated on this trial.

Participants may continue to receive magrolimab for up to 12 months or longer from the time of study entry, pending discussion with study chairs and study sponsor. Participants will be followed for up to 5 years after completion of treatment, or until removal from study, or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

Study Participants in Stratum A and Stratum B:

* Diagnosis of recurrent or progressive malignant primary brain tumor (WHO grade III or IV), including recurrent ependymoma (WHO grade II and III).
* Histologic confirmation of malignancy at original diagnosis or relapse is required for study entry.
* Participants must have measureable disease. Measurable disease will be defined as lesions that can be accurately measured in two dimensions (longest diameters to be recorded) with a minimum size of no less than double the slice thickness. Previously irradiated lesions are considered non-measurable except in cases of documented progression of the lesion since the completion of radiation therapy.
* Prior Therapy:

  * The patient must have failed at least one prior therapy, with or without surgery, prior to study registration. Prior therapies may include one of more of the following interventions: chemotherapy, immunotherapy, radiotherapy. Surgery alone does not constitute prior therapy. Patients must have fully recovered from clinically relevant acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
  * Myelosuppressive chemotherapy: Patients must have received their last dose of known myelosuppressive anticancer chemotherapy at least three weeks prior to study registration or at least six weeks prior if nitrosourea or mitomycin C.
  * Biologic agent: Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the biologic agent ≥ 7 days prior to study registration.
  * For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended to beyond the time during which adverse events are known to occur. The duration of this interval should be discussed with the study chair.
  * For biologic agents that have a prolonged half-life, the appropriate interval since last treatment should be discussed with the Study Chair prior to registration.
* Monoclonal antibody treatment: At least 28 days or 4 half-lives must have elapsed prior to registration, whichever is shorter. Such patients should be discussed with the study chair prior to registration.
* Bone Marrow Transplant:

  o Patients must be >= 3 months since autologous bone marrow/stem cell prior to registration
* Radiation:

  * Participants must have:
  * Had their last fraction of local irradiation to primary tumor >=12 weeks prior to registration; investigators are reminded to review potentially eligible cases to avoid confusion with pseudo-progression.
  * Had their last fraction of craniospinal irradiation or total body irradiation >+ 12 weeks prior to registration.
  * Had their last fraction of palliative radiation ≥ 14 days prior to registration.
* Performance Score: Karnofsky >= 50 for participants > 16 years of age and Lansky >=50 for participants <=16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Corticosteroids:

  o Participants who are receiving corticosteroids must be on a stable or decreasing dose for at least 7 days prior to enrollment. Stable dose should not be greater than dexamethasone 0.1 mg/kg/day (maximum 4 mg/day) or equivalent dose of alternate corticosteroid (physiologic replacement only).
* Organ Function Requirements:

  * Adequate Bone Marrow Function Defined as:

    * Peripheral absolute neutrophil count (ANC) 1000 mm3.
    * Platelet count 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
    * Hemoglobin>= 9.5 g/dL (RBC transfusions are permitted during the Screening Period and prior to enrollment to meet the hemoglobin inclusion criteria)
  * Adequate Renal Function Defined as:

    * Creatinine clearance or radioisotope Glomerular filtration rate (GFR) >= 60 millilitre (mL) per minute (mL/min) 1.73 m2 or
    * A serum creatinine based on age/gender as follows:
  * Age: 2 to < 6 years, Maximum Serum Creatinine (mg/dL): Male 0.8, Female 0.8.
  * Age: 6 to < 10 years, Maximum Serum Creatinine (mg/dL): Male 1.0, Female 1.0.
  * Age: 10 to < 13 years, Maximum Serum Creatinine (mg/dL): Male 1.2, Female 1.2.
  * Age: 13 to < 16 years, Maximum Serum Creatinine (mg/dL): Male 1.5, Female 1.4.
  * Age: >= 16 years, Maximum Serum Creatinine (mg/dL): Male 1.7, Female 1.4.
  * The threshold creatinine values in this table were derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the Center for Disease Control (CDC).
  * Adequate Liver Function Defined as:

    * Bilirubin (sum of conjugated + unconjugated) <= 1.5 x upper limit of normal (ULN) for age, or 3.0 x ULN and primarily unconjugated if patient has a documented history of Gilbert's syndrome or genetic equivalent. Institutions whose total bilirubin ULN is < 1.2 mg/dL may adopt 1.2 mg/dL as their ULN.
    * Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase ≤ 2.5x ULN.
    * Serum albumin ³ 2 g/dL.
* Adequate Neurologic Function Defined as:

  o Participants with seizure disorder may be enrolled if well controlled.
* The effects of magrolimab on the developing human fetus are unknown, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 4 months after completion of magrolimab administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* A legal parent/guardian or patient must be able to understand, and willing to sign, a written informed consent and assent document, as appropriate.

Exclusion Criteria:

* Participants who have had chemotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) or radiotherapy within 12 weeks prior to entering the study or those who have not recovered from clinically relevant acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
* Participants who are receiving any other investigational therapeutic agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to magrolimab, Ferumoxytol, or iron contained drugs or supplements.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active systemic infection.
* Women of childbearing potential must not be pregnant or breast-feeding.
* Participant has a known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Participant has any prior positive test result for hepatitis B virus or hepatitis C virus indicating presence of virus, e.g., hepatitis B surface antigen ((HBsAg), Australia antigen) positive, or hepatitis C antibody (anti-HCV) positive, except if HCV-RNA negative.
* Prior treatment with CD47 or SIRPα targeting agents.
* Prior hemolytic anemia or Evans Syndrome in the last 3 months.
* RBC transfusion dependence, defined as requiring more than 2 units of RBCs transfused during the 4-week period prior to screening. RBC transfusions are permitted during the screening period and prior to enrollment to meet the hemoglobin inclusion criteria. Participants who require three or more units of RBCs during the 4-week period prior to enrollment.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Participants with midline tumors, including midline HGG, DIPG, and diffuse midline glioma (DMG) or primary spinal cord tumors. Participants with disseminated disease are eligible.
* Participants at risk for imminent herniation, clinical evidence of significant increased intracranial pressure, or with >1 cm midline shift.
* Participants with a contraindication to MRI (metal implants).
* Participants with hemosiderosis/hemochromatosis, or iron overload from any cause (not just hemosiderosis or hemochromatosis), even if secondary to frequent blood transfusions, severe chronic hemolysis, excess dietary or parenteral iron, or any other etiology.
* Participants who have received a live vaccine within the last 30 days.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Up to 1 cycle (1 cycle is equal to 28 days)
  The investigator will employ the Bayesian optimal interval (BOIN) design to find the maximum tolerated dose (MTD). If the observed dose-limiting toxicity rate at the current dose is <= 0.236, the next cohort of patients will be treated at the next higher dose level; if it is >= 0.359, the next cohort of patients will be treated at the next lower dose level.
Proportion of participants with treatment-emergent adverse events | Up to 12 months
  The severity of toxicities will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Adverse events and will be summarized by maximum intensity and relationship to study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PhD, Principal Investigator — University of California, San Francisco; Nicholas Whipple, MD, MPH, Study Chair — University of Utah; Samuel Cheshier, MD, PhD, Study Chair — University of Utah; Howard Colman, MD PhD FAAN, Study Chair — University of Utah
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
De-identified, individual participant data may be shared with other researchers
Supporting Information: Study Protocol